CLINICAL TRIAL: NCT06588309
Title: What's in a Name? Do PTSD and Complex PTSD Diagnoses Predict Differences in Course and Outcome of Integrated Addiction and Trauma Focused Treatment?
Brief Title: The Course and Outcome of Integreated Trauma and Addiction Treatment Between PTSD and CPTSD
Status: Recruiting | Type: Observational
Sponsor: IrisZorg (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CPTSS
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: PTSD; Addiction
Keywords: PTSD; CPTSD; Addiction; EMDR; CRA
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Behavior, Addictive | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Addiction and PTSD
  Interventions: Behavioral: Eye movement desensitization and reprocessing (EMDR); Behavioral: CRA
- Addiction and CPTSD
  Interventions: Behavioral: Eye movement desensitization and reprocessing (EMDR); Behavioral: CRA

INTERVENTIONS:
Behavioral: Eye movement desensitization and reprocessing (EMDR) — Integrated addiction and traumafocused treatment.
Behavioral: CRA — CRA is a comprehensive cognitive behavioural treatment that focuses on helping people discover and adopt a pleasurable, social and healthy lifestyle that is more rewarding than a lifestyle including substance use.

SUMMARY:
In the ICD-11 post-traumatic stress disorder (PTSD) and complex PTSD (CPTSD) are distinguished. CPTSD is associated with early childhood traumatization and more severe symptom patterns. Research thus far confirms that PTSD and CPTSD are two related but different concepts, but it's still unclear what the clinical relevance of this differentiation is. In addiction care approximately one out of three patients suffer from (C)PTSD. It's unclear if in patients with a substance use disorder (SUD) comorbid CPTSD results in poorer treatment outcomes compared to comorbid PTSD.

DETAILED DESCRIPTION:
Rationale: In the ICD-11 post-traumatic stress disorder (PTSD) and complex PTSD (CPTSD) are distinguished. CPTSD is associated with early childhood traumatization and more severe symptom patterns. Research thus far confirms that PTSD and CPTSD are two related but different concepts, but it's still unclear what the clinical relevance of this differentiation is. In addiction care approximately one out of three patients suffer from (C)PTSD. It's unclear if in patients with a substance use disorder (SUD) comorbid CPTSD results in poorer treatment outcomes compared to comorbid PTSD.

Objective: To determine differences in course and outcome of integrated trauma-focused treatment delivered alongside addiction treatment in participants with comorbid PTSD and CPTSD.

Study design: An observational, prospective study with two groups (N = 50, allocation ratio 1:1) of participants with a SUD. One group has a comorbid PTSD (n = 25) and the other a comorbid CPTSD (n = 25). Assessments take place at baseline (T0), after every trauma- focused treatment session (T11-9) and after 10 weeks during which trauma-focused treatment may or may not have been completed or prematurely terminated (T2).

Study population: Patients with SUD and either comorbid PTSD or CPTSD, aged ≥ 18 years, with good Dutch language proficiency, who receive addiction treatment and trauma-focused treatment and who provide written informed consent.

Intervention: Treatment as usual (TAU), in accordance with the Dutch clinical practice guidelines consists of 1) addiction treatment according to the Community Reinforcement Approach (henceforth CRA) and 2) trauma-focused treatment (EMDR-therapy, henceforth EMDR).

Main study parameters/endpoints: Changes in PTSD symptom severity in participants with comorbid PTSD and CPTSD from T0 to T2, as measured by the PCL-5 and CAPS-5.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: All participants receive TAU, both CRA and EMDR, including standardized assessments. Additionally, participants fill in one extra questionnaire (ITQ) at T0 and T2 and the CAPS is administered additionally at T2. The extra burden of filling the ITQ is approximately one minute and for the CAPS approximately ten to forty-five minutes depending on the amount of symptoms after trauma treatment. Given the observational nature of the study, no risks related to the study are expected beyond those associated with routine clinical addiction care (e.g. relapse).

To optimize data-collection, especially after termination of EMDR before T2 assessment, participants receive an incentive, a voucher worth 10 euro, after completing the baseline (T0) assessment and the first five PCL-5 assessments (T11-5), and a voucher worth 15 euro after completing the next four PCL-5 assessments (T16-9) and the final assessment (T2).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years. •- Primary diagnosis SUD involving one of the following substances: alcohol, cannabis, cocaine, amphetamine, benzodiazepine, opioid according to the DSM-5 (American Psychiatric Association, 2013), who are receiving or starting outpatient CRA.

  * A DSM-5 diagnosis of PTSD (n=25). A DSM-5 diagnosis of PTSD and an additional ICD-11 diagnosis of CPTSD (n=25).
  * Planned start of EMDR-therapy within 8 weeks.
  * Good Dutch language proficiency (based on clinical judgement).
  * Written informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 50 eligible patients are enrolled from an outpatient treatment site of IrisZorg, a Dutch care provider for addiction care and sheltered housing. Patients will be screened at intake for addiction treatment. An additional screening can be performed during addiction treatment when symptoms of PTSD are suspected.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PTSD symptom severity | September 2023- September 2025
  Changes over time in PTSD symptom severity between participants with comorbid PTSD and CPTSD from T0-T2 as measured by the PCL-5.
Proportion of lost of the (C)PTSD diagnosis | September 2023- September 2025
  Proportion loss of (C)PTSD diagnoses in EMDR completers (as determined by their therapists) in both groups at end of treatment (T2) as measured by the ITQ and CAPS-5.

SECONDARY OUTCOMES:
substance use severity | September 2023- September 2025
  • Changes in substance use between participants with comorbid PTSD and CPTSD from T0 to T2, as measured by the MATE, section one

OTHER OUTCOMES:
(Serious) adverse events | September 2023- September 2025
  Occurrence of (serious) adverse events at T0 (past month) and during trauma treatment (T11-9).
  MDR treatment adherence: no-show and treatment drop-out.
EMDR treatment adherence | September 2023- September 2025
  number no-show and treatment drop-out during trauma focused treatment

CONTACTS AND LOCATIONS:
Locations (1):
- IrisZorg, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: No
Depending on the final data collection and the journal in which these are published, we will decide on availability of IPD